CLINICAL TRIAL: NCT05071404
Title: Efficacy Assessment and Monitoring of Subcutaneous Infliximab Levels in Patients With Inflammatory Bowel Disease.
Brief Title: Efficacy Assessment and Monitoring of Subcutaneous Infliximab Levels.
Acronym: Infliximab
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-INF-2020-01
Record Dates: First submitted 2021-09-16; First posted 2021-10-08 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2020-10

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients treated with infliximab sc.

SUMMARY:
Retrospective observational study in which the efficacy of infliximab is studied in patients with inflammatory bowel disease and its subcutaneous levels are monitored.

DETAILED DESCRIPTION:
Retrospective observational study in which the efficacy of infliximab is studied in patients with inflammatory bowel disease and its subcutaneous levels are monitored.

Treatment is prior to and independent of the patient's participation in the study and is governed by clinical judgment criteria and routine clinical practice, not performing any diagnostic or follow-up intervention that is not routine clinical practice.

Patients are older than 14 years who suffer from inflammatory bowel disease and who receive remsima as routine treatment.

The source of information will be the patient's medical history.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease.
* Over 14 years old.
* Receive Remsin as a treatment for his disease. And always this treatment that the patient is going to receive is governed by the criteria of clinical judgment and routine clinical practice, not performing any diagnostic or follow-up intervention that is not routine clinical practice.

Exclusion Criteria:

* Patients with inflammatory bowel disease under 14 years of age.
* Or older than this age with inflammatory bowel disease who do not attend the established check-ups

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with inflammatory bowel disease over 14 years of age who are being treated with infliximan sc.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Perform an efficacy assessment and monitoring of subcutaneous infliximab levels in patients with inflammatory bowel disease. | Up to 16 weeks.
  Number of hospitalizations of patients treated with subcutaneous infliximab suffering from inflammatory bowel disease.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Arguelles Arias, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain